CLINICAL TRIAL: NCT01448226
Title: Diagnosing Invasive Aspergillosis by PCR Based Investigation of Bronchoalveolar Lavage Samples During Antifungal Therapy
Brief Title: Diagnosing Invasive Aspergillosis by Polymerase Chain Reaction (PCR) Based Investigation of Bronchoalveolar Lavage Samples During Antifungal Therapy
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dieter Buchheidt, Prof. Dr. med., Heidelberg University
Other Study IDs: Aspergillus PCR BAL Study
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Invasive Aspergillosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Aliquots of BAL Samples including fungal DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- proven or probable aspergillosis
- possible aspergillosis

SUMMARY:
Invasive pulmonary aspergillosis (IPA) remains a major cause for morbidity and mortality in patients (pts) with hematologic malignancies. As culture-based methods only yield results in a minority of patients, using non-culture-based methods for detection of aspergillosis in clinical specimens becomes increasingly important. Analyzing bronchoalveolar lavage (BAL) samples with polymerase chain reaction (PCR) is promising, however, the influence of current antifungal drugs on the performance of this diagnostic tool remains controversial.

The aim of the trial is to elucidate on the performance of BAL PCR under antifungal treatment.

DETAILED DESCRIPTION:
Invasive pulmonary aspergillosis (IPA) remains a major cause for morbidity and mortality in patients (pts) with hematologic malignancies. As culture-based methods only yield results in a minority of patients, using non-culture-based methods for detection of aspergillosis in clinical specimens becomes increasingly important. Analyzing bronchoalveolar lavage (BAL) samples with polymerase chain reaction (PCR) is promising, however, the influence of current antifungal drugs on the performance of this diagnostic tool remains controversial.

The aim of the trial is to elucidate on the performance of BAL PCR under antifungal treatment.

Patients with high risk of invasive aspergillosis and lung infiltrates are sampled via BAL, the sample is analyzed for fungal DNA by Apsergillus specific PCR. Clinical data including treatment data is assessed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* immunocomprimised patients with high risk of invasive aspergillosis and lung infiltrates
* informed consent

Exclusion Criteria:

* Children under the age of 5 years
* Informed consent not available

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: immunocomprimised patients with lung infiltrates and high risk for invasive aspergillosis
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2000-01; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Buchheidt, MD, Principal Investigator — Mannheim University Hospital
Locations (22):
- Innsbruck University Hospital, Innsbruck, Austria
- Germany (21):
  - Bielefeld evangelisches Krankenhaus, Bielefeld
  - Bochum University Hospital, Bochum
  - Cologne University Hospital, Cologne
  - Düsseldorf University Hospital, Düsseldorf
  - Erlangen University Hospital, Erlangen
  - St.-Antonius Hospital Eschweiler, Eschweiler
  - General Hospital Frankfurt (Oder), Frankfurt (Oder)
  - Freiburg University Hospital, Freiburg im Breisgau
  - Halle University Hospital, Halle
  - Heidelberg University Hospital, Heidelberg
  - Herne University Hospital, Herne
  - Bone Marrow Transplantation Centre Idar-Oberstein, Idar-Oberstein
  - Jena University Hospital, Jena
  - Ludwigshafen General Hospital, Ludwigshafen
  - Mannheim University Hospital, Mannheim
  - Passau General Hospital, Passau
  - Potsdam General Hospital Ernst-von-Bergmann, Potsdam
  - Rostock University Hospital, Rostock
  - Ulm University Hospital, Ulm
  - Bone Marrow Transplantation Centre Wiesbaden, Wiesbaden
  - Würzburg University Hospital, Würzburg

REFERENCES:
- [Background] Skladny H, Buchheidt D, Baust C, Krieg-Schneider F, Seifarth W, Leib-Mosch C, Hehlmann R. Specific detection of Aspergillus species in blood and bronchoalveolar lavage samples of immunocompromised patients by two-step PCR. J Clin Microbiol. 1999 Dec;37(12):3865-71. doi: 10.1128/JCM.37.12.3865-3871.1999. PMID 10565898
- [Background] Buchheidt D, Baust C, Skladny H, Ritter J, Suedhoff T, Baldus M, Seifarth W, Leib-Moesch C, Hehlmann R. Detection of Aspergillus species in blood and bronchoalveolar lavage samples from immunocompromised patients by means of 2-step polymerase chain reaction: clinical results. Clin Infect Dis. 2001 Aug 15;33(4):428-35. doi: 10.1086/321887. Epub 2001 Jul 6. PMID 11462176
- [Background] Spiess B, Buchheidt D, Baust C, Skladny H, Seifarth W, Zeilfelder U, Leib-Mosch C, Morz H, Hehlmann R. Development of a LightCycler PCR assay for detection and quantification of Aspergillus fumigatus DNA in clinical samples from neutropenic patients. J Clin Microbiol. 2003 May;41(5):1811-8. doi: 10.1128/JCM.41.5.1811-1818.2003. PMID 12734210
- [Background] Hummel M, Spiess B, Cornely OA, Dittmer M, Morz H, Buchheidt D. Aspergillus PCR testing: results from a prospective PCR study within the AmBiLoad trial. Eur J Haematol. 2010 Aug;85(2):164-9. doi: 10.1111/j.1600-0609.2010.01452.x. Epub 2010 Apr 1. PMID 20374275